CLINICAL TRIAL: NCT05204615
Title: Prospective Data Collection for SENSING-AI: A Precision Digital and Wearables Platform for the Early Diagnosis of Emotional and Physical Complications in Patients With Long COVID Through the Use of Artificial Intelligence
Brief Title: SENSING-AI Cohort for Long COVID Patients
Acronym: SENSING-AI
Status: Completed | Type: Observational
Sponsor: Adhera Health, Inc. (Industry)
Collaborators: Fundación Pública Andaluza para la gestión de la Investigación en Sevilla (Other); Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Responsible Party: Sponsor
Other Study IDs: SEN-0221
Record Dates: First submitted 2022-01-10; First posted 2022-01-24 (Actual); Last update posted 2023-01-05 (Actual); Status verified 2022-01

CONDITIONS: Post-acute COVID-19 Syndrome
Keywords: COVID-19 syndrome; Prospective study; Artificial Intelligence; Mental Health
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Psychological Well-Being | interventions — Psychometrics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Prospective Long COVID cases: The target population will be 10 patients diagnosed during 2021 with long COVID, who will then be followed-up for one month.
  Interventions: Other: Collection of clinical, psychometric and biometric data

INTERVENTIONS:
Other: Collection of clinical, psychometric and biometric data — Wearable devices and a mobile app will be used to collect real-time data for 4 weeks to detect physiological and psychological complications based on biometric and psychometric (patient-reported outcomes) information.

SUMMARY:
The prospective study will focus on the collection of biometric and psychometric data from a limited population for 1 month with the aim of complementing the SENSING-AI retrospective cohort.

DETAILED DESCRIPTION:
The stratification of the risk of complications related to persistent COVID symptoms both physiological and psychological in a personalized way would optimize the cost-effectiveness model for the management of these patients. Similarly, the early detection of complications associated with persistent COVID in patients belonging to vulnerable groups would improve care times and, therefore, the patient's prognosis.

The primary objective of this study is to complement the SENSING-AI cohort with biometric and psychometric data prospectively gathered from patients diagnosed with long COVID in the last year to drive the generation of AI-based risk prediction and stratification models.

ELIGIBILITY:
Inclusion Criteria:

* Legal adults
* With a long COVID-19 diagnose in the last year
* Reporting any of these symptoms:
* Fatigue
* Dyspnea
* Shortness of breath
* Anxiety
* Stress
* Depression
* Conduct disorder
* Sleep disorder

Exclusion Criteria:

* Hospital admission during follow-up due to pathology not related to COVID-19
* Patients without digital literacy or who cannot use the mobile application.
* Known severe psychiatric illness or cognitive impairment
* Being pregnant (or suspected to be pregnant)
* Discharged after hospital admission due to COVID-19

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Sample will be recruited from patients attending Primary Care Aljarafe-Sevilla Norte centers and Jordi Gol Primary Care Research Institute.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2022-01-18 (Actual); Primary Completion 2022-02-12 (Actual); Study Completion 2022-04-28 (Actual)

PRIMARY OUTCOMES:
Physical Activity Distances | 1 month
  Through the Withings Scanwatch the following physical activity data are gathered: Daily distance travelled in metres; List of distance travelled/ 4-5 minutes approx.; Daily number of floors climbed in metres; List of distance travelled/ approx. 4-5 minutes.
Physical Activity in Steps | 1 month
  Through the Withings Scanwatch the following physical activity data are gathered: Daily number of steps; List of steps/ 4-5 minutes approximately.
Physical Activity Duration | 1 month
  Through the Withings Scanwatch the following physical activity data are gathered: Daily duration of light, moderate and intense intensity activities in seconds; Daily sum of moderate and intense activities in seconds.
Physical Activity Kcal | 1 month
  Through the Withings Scanwatch the following physical activity data are gathered: Daily active calories burned in Kcal; Total daily calories burned in Kcal; List of calories burned/ approx. 4-5 minutes.
Physical Activity Bpm | 1 month
  Through the Withings Scanwatch the following physical activity data are gathered: Daily minimum/average/maximum heart rate in bpm.
Physical Activity Heart Rate | 1 month
  Through the Withings Scanwatch the following physical activity data are gathered: Daily duration in seconds of heart rate; List of heart rate measurements/10 minutes/average rate.
Physical Activity Oxygen Saturation | 1 month
  Through the Withings Scanwatch the following physical activity data are gathered: Manual Oxygen Saturation (SpO2) measurements.
Workouts Kcal | 1 month
  Through the Withings Scanwatch the following workouts data are gathered: Calories / workout events in Kcal.
Workouts distances | 1 month
  Through the Withings Scanwatch the following workouts data are gathered: Distance of the workouts in meters; Steps climbed in metres; Step run in meters.
Workouts Bpm | 1 month
  Through the Withings Scanwatch the following workouts data are gathered: Heart rate/minimum/average/maximum intensity in bpm.
Workouts Heart Rate | 1 month
  Through the Withings Scanwatch the following workouts data are gathered: Duration in the minimum/moderate/intense heart rate zone in seconds; Duration of maximum heart rate in seconds.
Sleep quality Number of Times Awake | 1 month
  Through the Withings Scanwatch the following sleep quality data are gathered: Number of times the user woke up; Number of times the user got out of bed during the night.
Sleep quality duration | 1 month
  Through the Withings Scanwatch the following sleep quality data are gathered: Total time spent in bed in seconds; Total time asleep in seconds; Time spent in bed before falling asleep in seconds; Time spent in bed after waking up in seconds; Time spent awake in bed after falling asleep for the first time during the night in seconds; Duration in light resting state in seconds; Duration in deep sleep state in seconds; Ratio of total sleep time/time spent in bed.
Sleep quality Rapid Eye Movement | 1 month
  Through the Withings Scanwatch the following sleep quality data are gathered: Rapid Eye Movement (REM) sleep phase count.
Sleep quality Bpm | 1 month
  Through the Withings Scanwatch the following sleep quality data are gathered: Average heart rate in bpm; Average minimum bpm rate.
Sleep quality Breathing | 1 month
  Through the Withings Scanwatch the following sleep quality data are gathered: Intensity of breathing disturbances.
Fatigue Assessment Scale | Weekly up to 1 month
  The Fatigue Assessment Scale is a unidimensional scale, consisting of 10-items measured on 5-point rating scale varies from 1 never to 5 always. Scores range from 10 to 50 with higher scores indicating greater fatigue.
Dyspnoea Index | Weekly up to 1 month
  Dyspnoea Index is a unidimensional scale, consisting of 10-items evaluated on a 0-4 Likert Scale (0= never; 1= almost never; 2= sometimes; 3= almost always; 4= always). Scores range from 0 to 40 and higher scores indicate greater dyspnea.
Generalized Anxiety Disorder 7-Item Scale | Weekly up to 1 month
  Generalized Anxiety Disorder 7-Item Scale consists of 7 items measured on 4-point rating scale varies from 0 (not at all) to 3 (nearly every day). Scores range from 0 to 21 with higher scores indicating higher anxiety levels.
Perceived Stress Scale | Weekly up to 1 month
  Perceived Stress Scale consists of 10 items measures on 4-point rating scale varies from 0 (never) to 4 (nearly every day). Scores range from 0 to 40 with higher scores indicating higher perceived stress.
Patient Health Questionnaire-9 | Weekly up to 1 month
  Patient Health Questionnaire-9 consists of 9 items measures on 4-point rating scale varies from 0 (never) to 3 (nearly every day). Scores range from 0 to 27 and higher scores indicate higher depression levels.
Oviedo Sleep Questionnaire | Weekly up to 1 month
  Oviedo Sleep Questionnaire consists of 15 items, 13 form the scale itself and two are descriptive items to provide the clinician with information on parasomnias and on the type and frequency of use of any type of sleep aid. The 13 items are grouped in 3 subscales: a) Subjective satisfaction with sleep: 1 item. Likert scale of satisfaction with 7 values ranging from 1 (very dissatisfied) to 7 (very satisfied); b) Insomnia: made up of 9 items to assess the nature of insomnia (difficulties in reconciling sleep, maintenance, early awakening, non-restorative sleep) and its repercussions on wakefulness (worry/tiredness/decreased functioning. Scored on a 5-value Likert scale (from 1 to 5) where the higher the score, the greater the severity; c) Hypersomnia: consisting of 3 items that assess daytime sleepiness and concern/decreased functioning for this reason. Scored on a 5-value Likert scale (from 1 to 5) where the higher the score, the greater the severity.

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - IDIAP Jordi Gol, Barcelona
  - Primary Care Aljarafe-Sevilla Norte, Seville

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Michielsen HJ, De Vries J, Van Heck GL. Psychometric qualities of a brief self-rated fatigue measure: The Fatigue Assessment Scale. J Psychosom Res. 2003 Apr;54(4):345-52. doi: 10.1016/s0022-3999(02)00392-6. PMID 12670612
- [Background] Gartner-Schmidt JL, Shembel AC, Zullo TG, Rosen CA. Development and validation of the Dyspnea Index (DI): a severity index for upper airway-related dyspnea. J Voice. 2014 Nov;28(6):775-82. doi: 10.1016/j.jvoice.2013.12.017. Epub 2014 Oct 12. PMID 25311596
- [Background] Remor E. Psychometric properties of a European Spanish version of the Perceived Stress Scale (PSS). Span J Psychol. 2006 May;9(1):86-93. doi: 10.1017/s1138741600006004. PMID 16673626
- [Background] Campo-Arias A, Pedrozo-Pupo JC, Cogollo-Milanes Z. [PHQ-9 in screening of major depressive episode among COVID-19 survivors]. Rev Colomb Psiquiatr (Engl Ed). 2021 Jul 2. doi: 10.1016/j.rcp.2021.06.004. Online ahead of print. No abstract available. Spanish. PMID 34230698
- [Background] Johnson SU, Ulvenes PG, Oktedalen T, Hoffart A. Psychometric Properties of the General Anxiety Disorder 7-Item (GAD-7) Scale in a Heterogeneous Psychiatric Sample. Front Psychol. 2019 Aug 6;10:1713. doi: 10.3389/fpsyg.2019.01713. eCollection 2019. PMID 31447721
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Paz Garcia-Portilla M, Saiz PA, Diaz-Mesa EM, Fonseca E, Arrojo M, Sierra P, Sarramea F, Sanchez E, Goikole JM, Balanza V, Benabarre A, Bobes J. Psychometric performance of the Oviedo Sleep Questionnaire in patients with severe mental disorder. Rev Psiquiatr Salud Ment. 2009 Oct;2(4):169-77. doi: 10.1016/S1888-9891(09)73235-5. Epub 2010 Jan 25. English, Spanish. PMID 23034346
- [Derived] Fuster-Casanovas A, Fernandez-Luque L, Nunez-Benjumea FJ, Moreno Conde A, Luque-Romero LG, Bilionis I, Rubio Escudero C, Chicchi Giglioli IA, Vidal-Alaball J. An Artificial Intelligence-Driven Digital Health Solution to Support Clinical Management of Patients With Long COVID-19: Protocol for a Prospective Multicenter Observational Study. JMIR Res Protoc. 2022 Oct 14;11(10):e37704. doi: 10.2196/37704. PMID 36166648
- See also: Withings Scanwatch — https://www.withings.com/de/en/scanwatch